CLINICAL TRIAL: NCT05262790
Title: The Difference of Grey Matter Volume Among the Patients of Schizophrenia
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: GMV-2013
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia; Neuroimaging; Cognitive Dysfunction
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PNS group: The patients with prominently negative symptoms (PNS) had a greater score on the negative than on the positive subscale of the PANSS, a negative symptoms score > 20, and at least one of items from PANSS negative symptoms scale ≥ 4 points
  Interventions: Other: This is not an intervention study
- PPS group: The patients with predominantly positive symptoms (PPS) had a greater score on the positive than on the negative subscale of the PANSS
  Interventions: Other: This is not an intervention study
- Control: Healthy control
  Interventions: Other: This is not an intervention study

INTERVENTIONS:
Other: This is not an intervention study
  Groups: PNS group
Other: This is not an intervention study
  Groups: PPS group
Other: This is not an intervention study
  Groups: Control

SUMMARY:
Schizophrenia is a heritable complex phenotype whose symptoms can be clustered into three domains: positive symptoms, negative symptoms and cognitive impairments. Constellations of negative symptoms in SCZ are composed of diminished motivation and pleasure, such as asociality, anhedonia, and avolition, or diminished expressivity such as blunted affect and alogia. Negative symptoms are associated with decreased quality of life and poor functional outcomes. Although antipsychotics are generally effective on positive symptoms, they are poorly effective on negative symptoms Currently, there are no licensed targeted medications for negative symptoms. In view of these problems, considerable interest in identifying new treatment targets for negative symptoms has grown over the past decade. Despite intense efforts in brain imaging that have opened new opportunities for addressing these issues, the neurobiological mechanism of negative symptoms remains unclear.

Structural brain measures from magnetic resonance imaging (MRI) are highly heritable and representatively have high reproducibility and low measurement error. Prior neuroimaging researches have consistently shown neuroanatomical abnormalities in the brains of individuals with SCZ, with the most robust and consistent group-level structural differences in widespread reduced volumes of hippocampal thalamus, amygdala and nucleus accumbens. SCZ have been associated with widespread structural brain abnormalities, but results from neuroimaging studies have been inconsistent.

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is a heritable complex phenotype whose symptoms can be clustered into three domains: positive symptoms, negative symptoms and cognitive impairments. Constellations of negative symptoms in SCZ are composed of diminished motivation and pleasure, such as asociality, anhedonia, and avolition, or diminished expressivity such as blunted affect and alogia. Negative symptoms are associated with decreased quality of life and poor functional outcomes. Although antipsychotics are generally effective on positive symptoms, they are poorly effective on negative symptoms Currently, there are no licensed targeted medications for negative symptoms. In view of these problems, considerable interest in identifying new treatment targets for negative symptoms has grown over the past decade. Despite intense efforts in brain imaging that have opened new opportunities for addressing these issues, the neurobiological mechanism of negative symptoms remains unclear.

Structural brain measures from magnetic resonance imaging (MRI) are highly heritable and representatively have high reproducibility and low measurement error. Prior neuroimaging researches have consistently shown neuroanatomical abnormalities in the brains of individuals with SCZ, with the most robust and consistent group-level structural differences in widespread reduced volumes of hippocampal thalamus, amygdala and nucleus accumbens. SCZ have been associated with widespread structural brain abnormalities, but results from neuroimaging studies have been inconsistent.

ELIGIBILITY:
Inclusion Criteria:

* All the patients satisfied the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-Ⅳ) diagnostic criteria for schizophrenia or schizophreniform disorder.
* Women and men
* 18 to 60 years of age
* Able and willing to provide written informed consent; and willing to commit to the study protocol
* Able to read, speak, and understand Chinese

Exclusion Criteria:

* (i) were <18 years or >60 years
* (ii) psychotic patients in unstable clinical condition (e.g., being aggressive and uncooperative)
* (iii) had major neurological or other psychiatric disorders, or significant medical condition including neurological disease, severe cardiovascular, hepatic, renal diseases
* (iv)had MRI abnormalities, or had MRI contraindications.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Study population will include individuals with psychotic disorders (schizophrenia or schizophreniform disorder) and healthy comparison participants(without personal or family history of psychotic disorders). Participants will be women and men, all races and ethnicities. Participants with schizophrenia/schizophreniform disorder will be aged 18-60 years.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
GMV difference among PNS, PPS and HC groups. | baseline
  PNS、PPS and HC will undergo Magnetic Resonance Imaging (MRI) at baseline. And the GMV of the three group was collected and analysed.1)The PNS patients showed longer duration, less positive symptoms, more severe PANSS-total symptoms and negative symptoms (all p values ≤ 0.001) than PPS. 2)compared with HC group, PPS group showed reduced GMV in the right orbital gyrus.
Identifying genes associated with GMV alterations in PNS. | baseline
  1)PLS1 weighted gene expression profile was positively correlated with PNS vs. HC GMV difference.2)The 2 overlapping genes (GRM7, RASSF7) exhibited significant negative correlations with regional GMV alterations in schizophrenia patients with predominantly negative symptoms.
PPI network construction and hub gene identification. | baseline
  1)PPI analysis of hub genes revealed a network consisting of 10 connected proteins and 33 edges, which is remarkably significantly higher than the expected 2 edges.2)PPI analysis revealed a network consisting of 461 connected proteins and 706 edges, which is remarkably significantly higher than the expected 621 edges

IPD SHARING:
Plan to Share IPD: No